CLINICAL TRIAL: NCT06376864
Title: A Pilot Study Investigating the Effects of a Classroom-based Physical Activity Intervention on Executive Function, Physical Activity and Sedentary Behaviour in 8-12-year-old Children
Brief Title: Physical Activity Intervention Effects on Executive Function, Physical Activity and Sedentary Behaviour in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Gao Yang, Associate Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RC- FNRA-IG /20-21/SOSC/01
Record Dates: First submitted 2024-02-28; First posted 2024-04-19 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Child Behavior
Keywords: physical activity; sedentary behaviour; executive fundtion; health promotion; children
MeSH Terms: conditions — Child Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Activity Breaks intervention (Experimental): The intervention arm will receive the Activity Breaks intervention.
  Interventions: Behavioral: Activity Breaks
- The control group (No Intervention): The control arm will continue to receive their normal instruction.

INTERVENTIONS:
Behavioral: Activity Breaks — The Activity Breaks intervention is a 5-minute Activity Breaks programme that allows classroom teachers of all ages and ability levels to lead simple movement activities within their classrooms, negating the need for additional personnel or space.
  Arms: Activity Breaks intervention

SUMMARY:
The current study aims to implement the Activity Breaks intervention and evaluate its effectiveness on outcome measures of executive function (EF), physical activity (PA), and sedentary behaviour (SB) in school children.

DETAILED DESCRIPTION:
In Hong Kong, as well as globally, children fail to meet the current physical activity recommendations of 60-minutes of moderate-to-vigorous physical activity (MVPA) per day. Childhood and adolescence are critical periods for developing favourable lifestyle behaviours that can continue into adulthood. Health-promoting interventions that target physical inactivity are vitally important. Researchers have repeatedly demonstrated that higher academic achievement and better attendance at school occurs among children who are more physically active, healthy and fit. To promote improvements in health and education, it is essential to recognize movement as assistive to establishing cognitive and social skills. The current study aims to implement the Activity Breaks intervention and evaluate its effectiveness on outcome measures of executive function (EF), physical activity (PA), and sedentary behaviour (SB) in school children. The Activity Breaks intervention is a 5-minute Activity Breaks programme that allows classroom teachers of all ages and ability levels to lead simple movement activities within their classrooms, negating the need for additional personnel or space. It is expected that the 5-minute Activity Breaks programme performed three times a day over 8 weeks will not only increases daily PA, but also decreases SB through interrupting prolonged sitting time. The Activity Breaks Programme also improves executive functioning among primary school-aged children.

This study will be a pilot clustered randomised controlled trial involving 8 primary schools in Hong Kong. One class from each school will be recruited from primaries 4-6 (8-11-year-old children) as our target population. Schools randomised into the intervention will receive the Activity Breaks Programme whereas schools assigned to the control group will continue to receive their normal daily instruction.

Data will be collected from all participants (intervention and control) at three time points: Time 1 (T1) (baseline), Time 2 (T2) (Post-intervention), and Time 3 (T3) (3-month follow-up). The following pupil measures will be captured at all time points: 1. EF; 2. PA levels and SB patterns using accelerometers; and 3. anthropometric measurements. Two measures will be conducted among teachers including teacher interviews and teacher fidelity checks conducted using log books. All analyses will be performed using IBM SPSS statistical programmes. Multi-level modelling regression analyses with repeated measures will be used to determine the effects of the intervention. A mixed-design ANOVA with time (pre, post and follow-up) as a within-subject variable and group (intervention and control) as a between-subjects variable will be conducted, while adjusting for age, gender and body mass index.

ELIGIBILITY:
Inclusion Criteria:

* School children in primary school (exclude private or special education schools), grades 4-6 (8-12 years old)
* children with parental consent.

Exclusion Criteria:

* Children with diagnosed behavioural or learning problems (e.g., attention-deficit hyperactivity disorder, ADHD)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Executive function | baseline, 8 weeks, and 20 weeks
  The Wisconsin Card Sorting Test (WCST): The computerized version of the WCST will be used to assess flexibility in decision making in this study. The number of total errors and perseverative errors and failure to maintain a set will be used as scores.
Psychological capacities | baseline, 8 weeks, and 20 weeks
  Stroop Task. A computerized modified Stroop task will be used to reflect inhibition skills that help individuals override a prepotent response in favour of an alternative response.
Working memory | baseline, 8 weeks, and 20 weeks
  Digit Span Backward: In this test, a participant will be presented with a series of digits to be repeated backwards.
Attention | baseline, 8 weeks, and 20 weeks
  Measures of child attention levels will be measured using the online version of d2-R test of attention. TN-E is a total performance score which gives a measure of the relationship between performance accuracy and speed. TN-E scores are defined as 50-60% bad, 60-70% medium, 70-85% normal and over 85% is good.

SECONDARY OUTCOMES:
Physical activity (min/week) | baseline, 8 weeks, and 20 weeks
  The ActiGraph GT3X+ monitor (ActiGraph LLC, Pensacola, FL, USA) will be used to measure physical activity levels.
Sedentary behavior (hour) | baseline, 8 weeks, and 20 weeks
  The ActiGraph GT3X+ monitor (ActiGraph LLC, Pensacola, FL, USA) will be used to measure sedentary behavior.
Body weight (kg) | baseline, 8 weeks, and 20 weeks
  Body weight will be measured in light clothing to the nearest 0.1 kg with a calibrated electronic scale.
Height (cm) | baseline, 8 weeks, and 20 weeks
  Height will be measured without shoes to the nearest 0.1 cm using a stadiometer in accordance with standard procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Julien S. BAKER, PhD, Study Chair — HKBU; Wendy Yajun HUANG, PhD, Study Director — Sport, Physical Education and Health/SOSC/HKBU
Locations (1):
- Department of Sport, Physical Education, and Health, Hong Kong Bapist University, Kowloon Tong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartholomew JB, Jowers EM. Physically active academic lessons in elementary children. Prev Med. 2011 Jun;52 Suppl 1(Suppl):S51-4. doi: 10.1016/j.ypmed.2011.01.017. Epub 2011 Jan 31. PMID 21281672
- [Background] Bates ME, Lemay EP Jr. The d2 Test of attention: construct validity and extensions in scoring techniques. J Int Neuropsychol Soc. 2004 May;10(3):392-400. doi: 10.1017/S135561770410307X. PMID 15147597
- [Background] Carlson JA, Engelberg JK, Cain KL, Conway TL, Mignano AM, Bonilla EA, Geremia C, Sallis JF. Implementing classroom physical activity breaks: Associations with student physical activity and classroom behavior. Prev Med. 2015 Dec;81:67-72. doi: 10.1016/j.ypmed.2015.08.006. Epub 2015 Aug 19. PMID 26297105
- [Background] Brooke HL, Atkin AJ, Corder K, Ekelund U, van Sluijs EM. Changes in time-segment specific physical activity between ages 10 and 14 years: A longitudinal observational study. J Sci Med Sport. 2016 Jan;19(1):29-34. doi: 10.1016/j.jsams.2014.10.003. Epub 2014 Oct 16. PMID 25459234
- [Background] Carson V, Hunter S, Kuzik N, Gray CE, Poitras VJ, Chaput JP, Saunders TJ, Katzmarzyk PT, Okely AD, Connor Gorber S, Kho ME, Sampson M, Lee H, Tremblay MS. Systematic review of sedentary behaviour and health indicators in school-aged children and youth: an update. Appl Physiol Nutr Metab. 2016 Jun;41(6 Suppl 3):S240-65. doi: 10.1139/apnm-2015-0630. PMID 27306432
- [Background] Carson V, Hunter S, Kuzik N, Wiebe SA, Spence JC, Friedman A, Tremblay MS, Slater L, Hinkley T. Systematic review of physical activity and cognitive development in early childhood. J Sci Med Sport. 2016 Jul;19(7):573-8. doi: 10.1016/j.jsams.2015.07.011. Epub 2015 Jul 10. PMID 26197943
- [Background] Chesham RA, Booth JN, Sweeney EL, Ryde GC, Gorely T, Brooks NE, Moran CN. The Daily Mile makes primary school children more active, less sedentary and improves their fitness and body composition: a quasi-experimental pilot study. BMC Med. 2018 May 10;16(1):64. doi: 10.1186/s12916-018-1049-z. PMID 29743076
- [Background] Cliff DP, Hesketh KD, Vella SA, Hinkley T, Tsiros MD, Ridgers ND, Carver A, Veitch J, Parrish AM, Hardy LL, Plotnikoff RC, Okely AD, Salmon J, Lubans DR. Objectively measured sedentary behaviour and health and development in children and adolescents: systematic review and meta-analysis. Obes Rev. 2016 Apr;17(4):330-44. doi: 10.1111/obr.12371. Epub 2016 Feb 24. PMID 26914664
- [Background] Cole TJ, Bellizzi MC, Flegal KM, Dietz WH. Establishing a standard definition for child overweight and obesity worldwide: international survey. BMJ. 2000 May 6;320(7244):1240-3. doi: 10.1136/bmj.320.7244.1240. PMID 10797032
- [Background] Drummy C, Murtagh EM, McKee DP, Breslin G, Davison GW, Murphy MH. The effect of a classroom activity break on physical activity levels and adiposity in primary school children. J Paediatr Child Health. 2016 Jul;52(7):745-9. doi: 10.1111/jpc.13182. Epub 2016 May 11. PMID 27168479
- [Background] Dumith SC, Gigante DP, Domingues MR, Kohl HW 3rd. Physical activity change during adolescence: a systematic review and a pooled analysis. Int J Epidemiol. 2011 Jun;40(3):685-98. doi: 10.1093/ije/dyq272. Epub 2011 Jan 18. PMID 21245072
- [Background] Dunn LL, Venturanza JA, Walsh RJ, Nonas CA. An observational evaluation of move-to-improve, a classroom-based physical activity program, New York City schools, 2010. Prev Chronic Dis. 2012;9:E146. doi: 10.5888/pcd9.120072. PMID 22974754
- [Background] Fairclough SJ, Hackett AF, Davies IG, Gobbi R, Mackintosh KA, Warburton GL, Stratton G, van Sluijs EM, Boddy LM. Promoting healthy weight in primary school children through physical activity and nutrition education: a pragmatic evaluation of the CHANGE! randomised intervention study. BMC Public Health. 2013 Jul 2;13:626. doi: 10.1186/1471-2458-13-626. PMID 23819701
- [Background] Huang WY, Wong SHS, Sit CHP, Wong MCS, Sum RKW, Wong SWS, Yu JJ. Results from the Hong Kong's 2018 report card on physical activity for children and youth. J Exerc Sci Fit. 2019 Jan;17(1):14-19. doi: 10.1016/j.jesf.2018.10.003. Epub 2018 Oct 8. PMID 30662509
- [Background] Kobel, S., Kettner, S., Dreyhaupt, J., & Steinacker, J. M. (2017). Objectively Determined Physical Activity Levels in German Primary School Children after a One Year School-based Health Promoting Intervention. Journal of Childhood Obesity, 2 (2).
- [Background] Lavelle HV, Mackay DF, Pell JP. Systematic review and meta-analysis of school-based interventions to reduce body mass index. J Public Health (Oxf). 2012 Aug;34(3):360-9. doi: 10.1093/pubmed/fdr116. Epub 2012 Jan 20. PMID 22267291
- [Background] Lorentzen C, Ommundsen Y, Jenum AK, Holme I. The "Romsas in Motion" community intervention: program exposure and psychosocial mediated relationships to change in stages of change in physical activity. Int J Behav Nutr Phys Act. 2007 Apr 30;4:15. doi: 10.1186/1479-5868-4-15. PMID 17466077
- [Background] McMichan L, Gibson AM, Rowe DA. Classroom-Based Physical Activity and Sedentary Behavior Interventions in Adolescents: A Systematic Review and Meta-Analysis. J Phys Act Health. 2018 May 1;15(5):383-393. doi: 10.1123/jpah.2017-0087. Epub 2018 Mar 23. PMID 29570032
- [Background] Mahar MT, Murphy SK, Rowe DA, Golden J, Shields AT, Raedeke TD. Effects of a classroom-based program on physical activity and on-task behavior. Med Sci Sports Exerc. 2006 Dec;38(12):2086-94. doi: 10.1249/01.mss.0000235359.16685.a3. PMID 17146314
- [Background] Markland, D., & Tobin, V. (2004). A Modification to the Behavioural Regulation in Exercise Questionnaire to Include an Assessment of Amotivation. Journal of Sport and Exercise Psychology, 26(2), 191-196.
- [Background] Mullins NM, Michaliszyn SF, Kelly-Miller N, Groll L. Elementary school classroom physical activity breaks: student, teacher, and facilitator perspectives. Adv Physiol Educ. 2019 Jun 1;43(2):140-148. doi: 10.1152/advan.00002.2019. PMID 30933539
- [Background] Murtagh E, Mulvihill M, Markey O. Bizzy Break! The effect of a classroom-based activity break on in-school physical activity levels of primary school children. Pediatr Exerc Sci. 2013 May;25(2):300-7. doi: 10.1123/pes.25.2.300. Epub 2013 Mar 15. PMID 23504941
- [Background] Norris E, Dunsmuir S, Duke-Williams O, Stamatakis E, Shelton N. Protocol for the 'Virtual Traveller' cluster-randomised controlled trial: a behaviour change intervention to increase physical activity in primary-school Maths and English lessons. BMJ Open. 2016 Jun 27;6(6):e011982. doi: 10.1136/bmjopen-2016-011982. PMID 27354084
- [Background] Ridgers ND, Timperio A, Cerin E, Salmon J. Within- and between-day associations between children's sitting and physical activity time. BMC Public Health. 2015 Sep 23;15:950. doi: 10.1186/s12889-015-2291-3. PMID 26400793
- [Background] Routen, A. C., Johnston, J. P., Glazebrook, C., & Sherar, L. B. (2018). Teacher perceptions on the delivery and implementation of movement integration strategies: The CLASS PAL (Physically Active Learning) Programme. International Journal of Educational Research, 88, 48-59.
- [Background] Salmon J, Arundell L, Hume C, Brown H, Hesketh K, Dunstan DW, Daly RM, Pearson N, Cerin E, Moodie M, Sheppard L, Ball K, Bagley S, Paw MC, Crawford D. A cluster-randomized controlled trial to reduce sedentary behavior and promote physical activity and health of 8-9 year olds: the Transform-Us! study. BMC Public Health. 2011 Oct 4;11:759. doi: 10.1186/1471-2458-11-759. PMID 21970511
- [Background] Skrade, M. A. B. (n.d.). Integrated classroom physical activity: Examining perceived need satisfaction and academic performance in children p.93.
- [Background] Steele RM, van Sluijs EM, Sharp SJ, Landsbaugh JR, Ekelund U, Griffin SJ. An investigation of patterns of children's sedentary and vigorous physical activity throughout the week. Int J Behav Nutr Phys Act. 2010 Dec 9;7:88. doi: 10.1186/1479-5868-7-88. PMID 21143901
- [Background] Stewart JA, Dennison DA, Kohl HW, Doyle JA. Exercise level and energy expenditure in the TAKE 10! in-class physical activity program. J Sch Health. 2004 Dec;74(10):397-400. doi: 10.1111/j.1746-1561.2004.tb06605.x. PMID 15724566
- [Background] van Stralen MM, Yildirim M, Wulp A, te Velde SJ, Verloigne M, Doessegger A, Androutsos O, Kovacs E, Brug J, Chinapaw MJ. Measured sedentary time and physical activity during the school day of European 10- to 12-year-old children: the ENERGY project. J Sci Med Sport. 2014 Mar;17(2):201-6. doi: 10.1016/j.jsams.2013.04.019. Epub 2013 May 24. PMID 23707474
- [Background] Tandon PS, Tovar A, Jayasuriya AT, Welker E, Schober DJ, Copeland K, Dev DA, Murriel AL, Amso D, Ward DS. The relationship between physical activity and diet and young children's cognitive development: A systematic review. Prev Med Rep. 2016 Apr 22;3:379-90. doi: 10.1016/j.pmedr.2016.04.003. eCollection 2016 Jun. PMID 27419040
- [Background] Taylor SL, Noonan RJ, Knowles ZR, Owen MB, McGrane B, Curry WB, Fairclough SJ. Evaluation of a Pilot School-Based Physical Activity Clustered Randomised Controlled Trial-Active Schools: Skelmersdale. Int J Environ Res Public Health. 2018 May 17;15(5):1011. doi: 10.3390/ijerph15051011. PMID 29772839
- [Background] Tremblay MS, Barnes JD, Gonzalez SA, Katzmarzyk PT, Onywera VO, Reilly JJ, Tomkinson GR; Global Matrix 2.0 Research Team. Global Matrix 2.0: Report Card Grades on the Physical Activity of Children and Youth Comparing 38 Countries. J Phys Act Health. 2016 Nov;13(11 Suppl 2):S343-S366. doi: 10.1123/jpah.2016-0594. PMID 27848745
- [Background] Tremblay MS, Carson V, Chaput JP, Connor Gorber S, Dinh T, Duggan M, Faulkner G, Gray CE, Gruber R, Janson K, Janssen I, Katzmarzyk PT, Kho ME, Latimer-Cheung AE, LeBlanc C, Okely AD, Olds T, Pate RR, Phillips A, Poitras VJ, Rodenburg S, Sampson M, Saunders TJ, Stone JA, Stratton G, Weiss SK, Zehr L. Canadian 24-Hour Movement Guidelines for Children and Youth: An Integration of Physical Activity, Sedentary Behaviour, and Sleep. Appl Physiol Nutr Metab. 2016 Jun;41(6 Suppl 3):S311-27. doi: 10.1139/apnm-2016-0151. PMID 27306437
- [Background] Tremblay MS, Gray CE, Akinroye K, Harrington DM, Katzmarzyk PT, Lambert EV, Liukkonen J, Maddison R, Ocansey RT, Onywera VO, Prista A, Reilly JJ, Rodriguez Martinez MP, Sarmiento Duenas OL, Standage M, Tomkinson G. Physical activity of children: a global matrix of grades comparing 15 countries. J Phys Act Health. 2014 May;11 Suppl 1:S113-25. doi: 10.1123/jpah.2014-0177. PMID 25426906
- [Background] Tremblay MS, LeBlanc AG, Kho ME, Saunders TJ, Larouche R, Colley RC, Goldfield G, Connor Gorber S. Systematic review of sedentary behaviour and health indicators in school-aged children and youth. Int J Behav Nutr Phys Act. 2011 Sep 21;8:98. doi: 10.1186/1479-5868-8-98. PMID 21936895
- [Background] Trost SG, Sallis JF, Pate RR, Freedson PS, Taylor WC, Dowda M. Evaluating a model of parental influence on youth physical activity. Am J Prev Med. 2003 Nov;25(4):277-82. doi: 10.1016/s0749-3797(03)00217-4. PMID 14580627
- [Background] Watson A, Timperio A, Brown H, Hesketh KD. A primary school active break programme (ACTI-BREAK): study protocol for a pilot cluster randomised controlled trial. Trials. 2017 Sep 19;18(1):433. doi: 10.1186/s13063-017-2163-5. PMID 28927442